CLINICAL TRIAL: NCT01155700
Title: A 24 Week, Open Label, Multi-center Evaluation of Pharmacokinetics and Pharmacodynamics, Efficacy and Safety of Omalizumab in Japanese Children (6 - 15 Years) With Inadequately Controlled Allergic Asthma Despite Current Recommended Treatment
Brief Title: Pharmacokinetics and Pharmacodynamics, Efficacy and Safety of Omalizumab in Japanese Children (6 - 15 Years)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIGE025B1301
Record Dates: First submitted 2010-06-30; First posted 2010-07-02 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Allergic Asthma
Keywords: omalizumab; allergic asthma; pediatric patients
MeSH Terms: interventions — Omalizumab

ARMS (1):
- Omalizumab (Experimental): Omalizumab treatment
  Interventions: Drug: omalizumab

INTERVENTIONS:
Drug: omalizumab

SUMMARY:
The primary purpose of this study is to examine whether the geometric mean of serum free IgE level at 24 weeks of the treatment period in Japanese pediatric patients (6 to 15 years of age) reaches under 25 ng/mL (target level). The investigators will also assess how well PK/PD data of Japanese children fit the global PK-PD modeling built from those of Caucasian adults and children, and assess efficacy and safety data in Japanese pediatric patients which will fulfill the Japanese health authority requirement for approval. Data obtained from the study is intended to be used to support the registration of pediatric indication of omalizumab in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Body weight and serum total IgE level within the dosing table range; body weight of 20 to 150 kg and serum total IgE levels of 30 to 1300 IU/mL
* Receiving asthma long-term control medications of high dose ICS (>200 µg/day FP or equivalent) and two or more controller medications out of LTRA, theophylline, sodium cromoglycate, LABA, or OCSs 12 weeks prior to the run-in period. These medications should be kept stable for 4 weeks prior to the run-in period and during the run-in period (except for management of asthma attacks/exacerbations)
* Having 2 or more asthma exacerbations requiring treatment with a doubling of the maintenance ICS dose for at least 3 days and/or systemic (oral or IV) corticosteroids in the past; one of these exacerbations must have occurred in the previous 12 months, which is documented in the medical record
* Demonstrating inadequately controlled asthma symptoms during the last 14 day run-in period based on the patient diary which meet any of the following:

Asthma symptoms every day; Night-time symptoms in ≥2 out of the last 14 days (missing data to be treated as a day with no symptoms); Limitation of daily activities in ≥2 out of the last 14 days (missing data to be treated as a day with no limitations)

Exclusion Criteria:

* With a history of food or drug related severe anaphylactoid or anaphylactic reaction(s)
* With positive skin reaction to the study drug at the run-in period
* With known hypersensitivity to any ingredients, including excipients (sucrose, histidine, polysorbate 20) of the study drug or drug related to omalizumab (e.g., monoclonal antibodies, polyclonal gamma globulin)
* With platelet level ≤ 100,000/µL (100 x 109/L) at the run-in period
* Who are taking intra-muscular depo-steroids within 4 weeks of the run-in period
* Who are taking systemic (oral or IV) corticosteroids for reasons other than asthma within 4 weeks of the run-in period (patients with chronic OCSs use for asthma are allowed)

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2010-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
To examine whether the geometric mean of serum free IgE level at 24 weeks of the treatment period in Japanese pediatric patients reaches under 25 ng/mL (target level). | 24 weeks

SECONDARY OUTCOMES:
To assess PK/PD data by modeling & simulation | 24 weeks
To assess the efficacy of omalizumab by PEF, pulmonary function, asthma symptom score, asthma rescue medication use and QOL questionnaire score. | 24 weeks
To assess the safety of omalizumab | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (15):
- Japan (15):
  - Novartis Investigative Site, Ohbu, Aichi-ken
  - Novartis Investigative Site, Chiba, Chiba
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Gifu, Gifu
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Tsu, Mie-ken
  - Novartis Investigative Site, Tenri, Nara
  - Novartis Investigative Site, Habikino, Osaka
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Shimotsuka-gun, Tochigi
  - Novartis Investigative Site, Fuchū, Tokyo
  - Novartis Investigative Site, Komae, Tokyo
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Sumida-ku, Tokyo

REFERENCES:
- [Result] Odajima H, Ebisawa M, Nagakura T, Fujisawa T, Akasawa A, Ito K, Doi S, Yamaguchi K, Katsunuma T, Kurihara K, Kondo N, Sugai K, Nambu M, Hoshioka A, Yoshihara S, Sato N, Seko N, Nishima S. Omalizumab in Japanese children with severe allergic asthma uncontrolled with standard therapy. Allergol Int. 2015 Oct;64(4):364-70. doi: 10.1016/j.alit.2015.05.006. Epub 2015 Jun 10. PMID 26433533